CLINICAL TRIAL: NCT00319475
Title: Evaluation of Mechanical Stapler for Aortic Anastomoses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SVSE 2000 Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-DE 006
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Aortic Aneurysm, Abdominal; Leriche Syndrome
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Leriche Syndrome

INTERVENTIONS:
Procedure: AAA or AF/IB (end-to-end) in patients with Leriche Syndrome

SUMMARY:
Demonstrate the safety and performance of the Aortic Stapler when used to attach a synthetic graft to an aorta in AAA and Leriche Syndrome patients

ELIGIBILITY:
Inclusion Criteria:

* Patient age is between 21 to 85 years old.
* Patient is diagnosed with Abdominal Aortic Aneurysm (AAA) or -aorto-Iliac/Femoral Occlusive Arterial Disease (Leriche' syndrome) by CT-Angio examination and/or angiography examination in patients with Leriche' syndrome.
* Patient with an aneurysm at the neck of the proximal or distal site that is between 5 to 10 mm and with a diameter of 16-22 mm.
* Patient is scheduled for AAA repair

Exclusion Criteria:

* Pregnant women
* Active malignancy
* Ruptured aneurysm
* Thoraco-AAA
* Patient with at least one of the following unstable risk factors:
* Renal disease (Cr >2)
* Ischemic heart disease (unstable Angina)
* Obstructive Pulmonary Disease (contraindicated for open aortic surgery by respiratory function exam)
* Severe CHF (EF < 25%)
* Patient with known allergy to metals or to the contrast media
* Participation in current or recent (within 60 days prior to surgery) clinical trial

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-02; Study Completion 2006-07

PRIMARY OUTCOMES:
Time to complete each stapled anastomosis.

SECONDARY OUTCOMES:
Post-operative follow up:
no leakage
no dilatation
no fistula or hematoma at the anastomotic sites

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kolvenbach, MD, Principal Investigator — Augusta Hospital, Berlin
Locations (1):
- Augusta Hospital, Düsseldorf, Germany